CLINICAL TRIAL: NCT05897138
Title: A Phase 2, Multi-Center, Single Arm Study to Evaluate Lenvatinib Plus Tislelizumab for Locally Advanced Unresectable or Metastatic Hepatocellular Carcinoma With Hepatitis B Virus Infection and Biomarker Analyses
Brief Title: A Study to Evaluate Lenvatinib Plus Tislelizumab for Locally Advanced Unresectable or Metastatic Hepatocellular Carcinoma With Hepatitis B Virus Infection and Biomarker Analyses
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Glitter-01
Record Dates: First submitted 2023-05-13; First posted 2023-06-09 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenvatinib plus Tislelizumab (Experimental)
  Interventions: Drug: Lenvatinib at a dose of 8 mg or 12 mg based on body weight + tislelizumab for one 21-day cycle

INTERVENTIONS:
Drug: Lenvatinib at a dose of 8 mg or 12 mg based on body weight + tislelizumab for one 21-day cycle — Drug: Lenvatinib Capsules administered orally once daily
  Drug: Tislelizumab 200 mg intravenous (IV) infusion administered on Day 1 of each cycle

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of Lenvatinib Plus Tislelizumab for Locally Advanced Unresectable or Metastatic Hepatocellular Carcinoma With Hepatitis B Virus Infection and Biomarker Analyses.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the efficacy and safety of Lenvatinib Plus Tislelizumab for Locally Advanced Unresectable or Metastatic Hepatocellular Carcinoma With Hepatitis B Virus Infection and Biomarker Analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent before screening;
2. Age ≤ 18 years old ≤75 years old for both men and women;
3. ECOG score 0-1;
4. A clinical or pathological diagnosis of hepatocellular carcinoma should meet one of the following criteria: ① A histological or cytological diagnosis of hepatocellular carcinoma, except for fibrolamellar, sarcomatoid or mixed cholangiocarcinoma; ② According to the Diagnosis and Treatment Guidelines for Primary Liver Cancer (2022 Edition), the patient was clinically diagnosed with HCC;
5. Hepatitis B virus surface antigen (HBsAg) positive and hepatitis B virus (HBV) DNA<2000IU/ml or 104 copies /ml; Or hepatitis B virus core antibody (HBcAb) positive, HBsAg negative, and highly sensitive HBV DNA<2000IU/ml or 104 copies /ml;
6. have not previously received any systemic therapy for HCC (mainly including systemic chemotherapy, antivascular therapy, molecular targeted therapy, immunotherapy targeting any other antibodies or drugs that act on T-cell co-stimulation or immune checkpoint pathways, Including but not limited to anti-PD-1, anti-PD-L1 /L2, anti-CD137 or anti-ctLA-4 antibodies), and disease progression 6 months after the end of postoperative adjuvant chemotherapy were allowed to be enrolled;
7. Chinese clinical stage of liver cancer (CNLC) Ⅲb or CNLC Ⅱb-Ⅲa which is not suitable for surgery and/or local treatment;
8. Child-Pugh rating for liver function: Grade A and good Grade B (≤7 points), and no history of hepatic encephalopathy;
9. There is at least one measurable lesion according to the efficacy evaluation criteria for solid tumors (RECIST version 1.1), and there is definite disease progression for lesions previously treated locally

Can be selected as a target lesion;

10) Expected survival of more than 3 months;

11) Major organ function is normal (no blood component, cell growth factor or albumin infusion therapy has been given within 14 days prior to laboratory examination), if the following criteria are met:

1. Blood routine: neutrophil ≥1.5×l09/L, platelet ≥75×109/L, hemoglobin ≥90g/L;
2. Liver function: alanine aminotransferase (ALT) and aspartate aminotransferase (AST), ALT and AST≤5×ULN; Serum albumin ≥28g/L; Total bilirubin (TBIL) ≤2×ULN; Alkaline phosphatase (ALP) ≤5×ULN;
3. Renal function: serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Ccr) ≥50mL/min;
4. Urine protein <2+ by routine detection; If urine protein ≥2+ at baseline, 24-hour urine protein quantity must be ≤1.0g;
5. Coagulation function: activated partial thromboplastin time (APTT), International Normalized Ratio (INR), prothrombin time (PT) ≤1.5×ULN;
6. Echocardiography: left ventricular ejection fraction (LVEF) ≥50%;

   Exclusion Criteria:
   1. Liver surgery and/or local treatment for HCC, except palliative radiotherapy for bone metastases to relieve pain, had been performed within 4 weeks prior to initial study drug therapy;
   2. Subjects (except hair loss and fatigue) who have not recovered from any toxicity and/or complications of local therapy (including interventional therapy, radio frequency therapy, etc.), previous chemotherapy, surgery, radiotherapy, that is, have not fallen to ≤ Grade 1 (NCI CTCAE version 5.0);
   3. Have received anti-tumor drug therapy in the past (including but not limited to traditional Chinese medicine preparations with anti-tumor indications);
   4. With moderate or severe ascites or ascites requiring drainage, or with pleural or pericardial effusion requiring drainage and/or symptoms of shortness of breath;
   5. with known active central nervous system metastases (CNS) and/or cancerous meningitis;
   6. With other malignancies (other than cured cervical carcinoma in situ, non-melanoma skin cancer or other tumors/cancers that have been treated radically and have shown no signs of disease for at least 5 years);

   (7) Combined history of bleeding tendency, high risk of bleeding, or cocoagulation dysfunction, including an arteriovenous thromboembolism event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, pulmonary embolism, deep vein thrombosis, or any other severe thromboembolism in the 6 months prior to screening;

   8) The portal vein cancer thrombus involved the main trunk, or both the main trunk and the superior mesenteric vein, or the inferior vena cava cancer thrombus or heart involvement;

   9) Unhealed wounds, active digestive tract ulcers or bleeding, fractures (excluding healed old fractures);

   10) Esophageal or gastric varicose bleeding occurred within 6 months prior to treatment, or severe varicose veins were known to exist on endoscopic examination.

   11) A history of gastrointestinal perforation and/or fistula, abdominal abscess, intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition), extensive enterectomy (partial resection of the colon or extensive resection of the small intestine with chronic diarrhea), Crohn's disease, ulcerative colitis, or long-term chronic diarrhea within 6 months prior to treatment;

   12) Patients who had undergone major surgery within 4 weeks prior to enrollment or expected to undergo major surgery during the study period (except for diagnostic biopsy);

   13) Having a known or suspected autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, autoimmune thyroid disease, multiple sclerosis, vasculitis, glomerulonephritis, etc.), having a history of human immunodeficiency virus infection (HIV positive), or having other acquired or congenital immunodeficiency diseases.

   14) Patients with a history of active tuberculosis or active or uncontrolled infection requiring systematic treatment (except simple urinary tract infection or upper respiratory tract infection) or syphilis infection requiring treatment;

   15) Subjects with a combined history of interstitial lung disease, non-infectious pneumonia, or high suspicion of having interstitial lung disease; Subjects with a history of drug-induced or radiological noninfectious pneumonia without symptoms were admitted;

   16) A history of severe medical disease, such as grade III or higher cardiac dysfunction (New York Heart Association [NYHA]), ischemic heart disease (such as myocardial infarction or angina), or myocardial infarction within the 3 months prior to enrollment, Subjects with poorly controlled diabetes (fasting blood glucose ≥10mmol/L) after medication or hypertension (systolic blood pressure >140mmHg and/or diastolic blood pressure >90mmHg) after medication and with prior hypertensive crisis or hypertensive encephalopathy;

   17) Receive live vaccines (except seasonal influenza vaccines that do not contain live viruses) within 4 weeks before the first study drug treatment or during the planned study period;

   18) Allergic to any component of tirelizumab or Lenvatinib, or known allergic to any other monoclonal antibody;

   19) Pregnant or lactating women, or subjects who plan to become pregnant during the treatment period and within 6 months after the end of treatment; Unwillingness to use effective contraception (including male subjects with the ability to impregnate women and female subjects and their male partners) during the study and for at least 6 months after the last study medication;

   20) The subject is known to have a history of drug addiction or mental illness;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | 12 months
  the proportion of participants who got a complete response (CR) and partial response (PR) according to RECIST v1.1.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | from first dose to within 30 days after the last dose
  Incidence of Treatment-Emergent Adverse Events were evaluated in accordance with the NCI CTC AE Version 5.0
Duration of response (DOR) | time from CR or PR (RECIST v1.1) achievement with investigational therapy, until documented progression, relapse, or death due to disease progression
  time from CR or PR (RECIST v1.1) achievement with investigational therapy, until documented progression, relapse, or death due to disease progression
Disease Control Rate (DCR) | 12 months
  the percentage of patients who have achieved CR, PR, and SD.
Progression-Free Survival (PFS) | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  the period from treatment initiation until the date of disease progression, death, or study cutoff, whichever occurred first.
Overall survival(OS) | From date of treatment until the date of death from any cause, whichever came first, assessed up to 100 months
  OS was defined as the time from the date of treatment to the date of death due to any cause. For subjects who were alive or lost to follow-up by the data analysis cut-off date, survival was censored at the subject's last known survival time.